CLINICAL TRIAL: NCT06782308
Title: Tinnitus Patient Preferences Survey
Status: Recruiting | Type: Observational
Sponsor: Nicolas Gninenko (Industry)
Responsible Party: Sponsor-Investigator, Nicolas Gninenko, Clinical Neuroscientist, Neurosoft Bioelectronics SA
Organization: Neurosoft Bioelectronics SA (Industry)
Other Study IDs: TEP-03301
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Tinnitus, Subjective; Tinnitus, Bilateral; Tinnitus, Noise Induced; Tinnitus, Hearing Loss, Cochlear Implant Users
Keywords: tinnitus; iBCI; brain implant; survey; risks acceptance; user preferences; patient preferences; subjective tinnitus; chronic tinnitus; severe tinnitus; catastrophic tinnitus; invasive neuromodulation; surgical treatment
MeSH Terms: conditions — Tinnitus; Hearing Loss; Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with tinnitus
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — patients preferences survey

SUMMARY:
The goal of this survey is to assess several aspects related to patient preferences regarding interventions for alleviating tinnitus through invasive electrical brain stimulation (neuromodulation). This survey covers the acceptance of a surgically-placed brain implant, of its associated risks related to the neurosurgical procedure, usability considerations, and the willingness/ability to pay for such a treatment.

Neurosoft Bioelectronics will use the collected patients' feedback and usability preferences data for the development of a novel minimally invasive brain implant aimed at alleviating tinnitus.

DETAILED DESCRIPTION:
Neurosoft Bioelectronics is developing a minimally invasive implantable solution for the treatment of chronic, subjective moderate-to-severe cases of tinnitus. The approach involves developing a state-of-the-art neurostimulation paradigm and incorporating invasive neuromodulation findings from leading experts in the field to create an effective solution. This solution aims to minimize patient's burden by offering a fully implantable system that does not require active patient engagement or repetitive adjustments of electrical stimulation parameters. Instead, it will use a closed-loop feedback algorithm, that will be optimized through multi-target recordings and stimulation, to continuously adapt and refine the treatment. This type of solution could significantly increase the quality of life of affected individuals living with severe chronic tinnitus, for which only palliative and symptom management solutions exist today. As Neurosoft Bioelectronics is at the early stage of device development, we will use the collected patients' feedback and usability preferences data for refining clear users' and product's requirements.

ELIGIBILITY:
Inclusion criteria:

* Individuals aged 18 or older suffering from subjective tinnitus
* Self-reported or healthcare professional-diagnosed chronic (lasting 3 months or longer), subjective, burdensome tinnitus

Exclusion criteria:

* Individuals under 18 years of age
* Healthy volunteers without tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (over 18 years old) with chronic, subjective severe tinnitus
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance of invasive neuromodulation treatments for chronic tinnitus | 1 year
  Risks acceptance and user preferences will be assessed through responses to the survey. The outcome will be summarized in the form of a percentage or similar statistics on acceptances rates for surgical interventions in patients with chronic tinnitus. Acceptance rates will also be evaluated in accordance to several clinical characteristics of tinnitus, such as its perceived annoyance or loudness.

SECONDARY OUTCOMES:
Usability preferences for implantable neuromodulation systems for chronic tinnitus | 1 year
  Usability preferences will be assessed through responses to the survey. This secondary outcome will be summarized in the form of a percentage or similar statistics on usability preferences between different solutions involving surgical interventions in patients with chronic tinnitus. Usability preferences will also be evaluated with respect to different reported tinnitus characteristics, such as perceived annoyance or loudness.
Willingness and ability to pay for novel invasive neuromodulation solutions for chronic tinnitus | 1 year
  Willingness to pay (WTP) will be assessed through responses to the survey. This secondary outcome will be summarized in the form of a range ($ US) or similar statistics on willingness and ability to pay with respect to different solutions involving surgical interventions in patients with chronic tinnitus. WTP will also be evaluated with respect to different reported tinnitus characteristics, such as perceived annoyance or loudness.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Gninenko, PhD, Principal Investigator — Neurosoft Bioelectronics
Locations (1):
- Neurosoft Bielectronics US Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.neurosoft-bio.com/tinnitus
- See also: Link to access the survey — https://survey.sogolytics.com/r/feCz2L